CLINICAL TRIAL: NCT04155983
Title: Ultrasound Guided Adductor Canal Block vs Intra-Operative Trans-Articular Saphenous Nerve Block: A Prospective Trial
Brief Title: High Versus Low Adductor Canal Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carilion Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-19-643
Record Dates: First submitted 2019-11-04; First posted 2019-11-07 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Osteo Arthritis Knee
Keywords: gonarthrosis; osteoarthritis; knee; total knee arthroplasty; adductor canal block; saphenous nerve block; multimodal pain control
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Study Design: Prospective RCT
  Study Groups:
  US Guided, Anesthesia Administered Adductor Canal Block ("High ACB") Intra-Operative, Surgeon Administered Adductor Canal Block ("Low ACB")
  Model- Cluster Randomization There will be two surgeons collecting data for this study; Dr. Mann (principal investigator) & Dr. Moskal. Each surgeon will begin collecting data on opposite arms of the study. Surgeon A will perform 35 consecutive High-ACB knees while Surgeon B performs 35 Low-ACB knees. After performing 35 knees under either the High-ACB or Low-ACB protocol, Surgeon A and Surgeon B will switch arms and perform an additional 35 consecutive knees in the opposite arm. At trial's end, each surgeon will have performed 35 TKAs using the High-ACB and Low-ACB protocol yielding a total of 70 patients in each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High ACB (Active Comparator): In the pre-operative cohort, the adductor canal block is administered by anesthesia staff immediately prior to patient transport to the operating room. The thigh is prepped with cholorhexidine at the midpoint between the anterior superior iliac spine and the patella and sterile drapes are applied. An ultrasound probe is then used to localize the adductor canal and confirm that the femoral artery, femoral vein and saphenous nerve can be visualized deep to the sartorious. The probe is moved proximally or distally until the neurovascular bundle is centered under the sartorius. A 20cc syringe with a blunt tip 1.5in 18ga needle is then used to inject 15cc of 0.5% ropivocaine. Following this, the wound is prepped and draped in usual sterile fashion for the arthroplasty procedure.
  Interventions: Drug: Ropivacaine
- Low ACB (Active Comparator): Surgeon Administered Group In the intra-operative cohort, the block will be administered after the final components are in place and cement debris is removed. The knee joint is irrigated with dilute hibiclens or betadine followed by pulsatile lavage per institutional protocol. A blunt tip 1.5in 18ga needle was then used to administer 15cc of 0.5% ropivocaine.. The location of the saphenous nerve as it exits the adductor canal will be estimated to be 1.5x the TEA proximal to the medial epicondyle in men and 1.3x the TEA proximal in women as described by Kavolus et al. The 60cc of the anesthetic will then injected through the vastus medialis musculature in a field extending from 1cm proximal to one cm distal to the assumed location of the nerve with the needle directed in from 20° to 45° medial. The wound is then irrigated pulsatile lavage one final time and closed in layered fashion.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — The drug will be administered in the same dosage in both arms. The location of the injection will vary by arm.
  Other Names: naropin

SUMMARY:
The investigators will be comparing the efficacy of two different techniques for performing an adductor canal block to the saphenous nerve as a part of the multimodal pain control regimen for total knee arthroplasty. The investigators will be comparing a "low adductor canal block" in which the surgeon administers local anesthetic to the distal aspect of the nerve from the operative site to a "high adductor canal block" in which the anesthesiologist administers the local anesthetic more proximally along the thigh using ultrasound guidance. The investigators will power the study for non-inferiority to compare the newer "low" block to the more commonly performed and more widely studied "high" block.

DETAILED DESCRIPTION:
Study Design: Prospective RCT

Study Question- Does a surgeon administered intra-operative adductor canal block ("Low-ACB") provide non-inferior post-operative pain relief relative to anesthesia administered, ultrasound guided adductor canal block ("High-ACB").

Hypothesis- Surgeon administered Low-ACB provides non-inferior pain relief relative to anesthesia administered High-ACB.

Study Groups-

1. US Guided, Anesthesia Administered Adductor Canal Block ("High ACB")
2. Intra-Operative, Surgeon Administered Adductor Canal Block ("Low ACB")

Randomization- Cluster Randomization There will be two surgeons collecting data for this study; Surgeon A (principal investigator) & Surgeon B. Each surgeon will begin collecting data on opposite arms of the study. Surgeon A will perform 35 consecutive High-ACB knees while Surgeon B performs 35 Low-ACB knees. After performing 35 knees under either the High-ACB or Low-ACB protocol, Surgeon A and Surgeon B will switch arms and perform an additional 35 consecutive knees in the opposite arm. At trial's end, each surgeon will have performed 35 TKAs using the High-ACB and Low-ACB protocol yielding a total of 70 patients in each arm.

Participant Timeline:

The investigators will interact with patients and collect specific data at a limited number of office visits as outlined below. All office appointments will take place at the Carilion Clinic Institute for Orthopaedics and Neurosciences.

1. Pre-Op Appointment- Thorough informed consent will be obtained at this visit. Patient will be sent home with consent form to review further and discuss with family.
2. Day of Surgery- Prior to surgery, operative team will go over consent one final time and obtain signature if patient consents.
3. Post-Op Admission- Standard post-op protocol will be followed. Data will be collected from this admission from the Epic EMR as above.
4. Discharge Home- Patient will keep pill journal for opioid narcotics taken each day as well as a recording their daily pain score prior to bed.
5. 2 Week F/U Appointment- PROMIS, KOOS Jr. and VAS scores as well as physical exam data recorded. This requires no additional time as this is part of routine post TKA follow up.
6. Home 2-6 Weeks- Patient will keep pill journal for opioid narcotics taken each day as well as a recording their daily pain score prior to bed.
7. 6 Week F/U Appointment- PROMIS, KOOS Jr. and VAS scores as well as physical exam data recorded. This requires no additional time as this is part of routine post TKA follow up.

At this point, the patient has completed their participation in the study and will continue follow up as scheduled without further data collection.

Technical Details:

Surgeon Administered Group In the intra-operative cohort, the block will be administered after the final components are in place and cement debris is removed. The knee joint is irrigated with dilute hibiclens or betadine followed by pulsatile lavage per institutional protocol. A A blunt tip 1.5in 18ga needle was then used to administer 15cc of 0.5% ropivocaine.. The location of the saphenous nerve as it exits the adductor canal will be estimated to be 1.5x the TEA proximal to the medial epicondyle in men and 1.3x the TEA proximal in women as described by Kavolus et al.[3] The 60cc of the anesthetic will then injected through the vastus medialis musculature in a field extending from 1cm proximal to one cm distal to the assumed location of the nerve with the needle directed in from 20° to 45° medial. The wound is then irrigated pulsatile lavage one final time and closed in layered fashion.

Anesthesia Administered Group In the pre-operative cohort, the adductor canal block is administered by anesthesia staff immediately prior to patient transport to the operating room. The thigh is prepped with cholorhexidine at the midpoint between the anterior superior iliac spine and the patella and sterile drapes are applied. An ultrasound probe is then used to localize the adductor canal and confirm that the femoral artery, femoral vein and saphenous nerve can be visualized deep to the sartorious. The probe is moved proximally or distally until the neurovascular bundle is centered under the sartorius. A 20cc syringe with a blunt tip 1.5in 18ga needle is then used to inject 15cc of 0.5% ropivocaine. Following this, the wound is prepped and draped in usual sterile fashion for the arthroplasty procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing unilateral primary TKA for primary osteoarthritis
* Age over 18

Exclusion Criteria:

* Pre-operative narcotic use
* Bilateral procedure
* Non-Primary arthroplasty
* Workman's comp
* Inability to have spinal anesthesia (blood thinners)
* Unsuccessful spinal anesthesia
* Inflammatory or Post Traumatic arthritis
* ASA score of 4
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Narcotic Consumption | Up to 48 hours after surgery
  Post-operative narcotic utilization measured in Morphine Equivalents per hour.
Narcotic Consumption | through study completion, an average of 6 weeks
  Post-operative narcotic utilization measured in Morphine Equivalents per hour.

SECONDARY OUTCOMES:
Length of stay | through study completion, an average of 6 weeks
  Length of hospital stay after surgery measured in hours
Visual Analog Scale Pain Scores | Recorded hourly while in hospital, daily after discharge up until 6wks
  10 point validated patient reported pain scores with 0 being no pain and 10 being the worst pain the patient can imagine.
Inpatient therapy | Up to 48 hours after surgery
  Number of steps taken at each therapy session while in the hospital
Patient Reported Outcome Measure Information System 10 Score | through study completion, an average of 6 weeks
  validated outcome measure using 10 questions and scored on a 50 point scale with 0 being the worst and 50 being the best overall score.
Knee injury and Osteoarthritis Outcome Score Junior | through study completion, an average of 6 weeks
  validated outcome measure using 7 questions and scored on a 100 point scale such that 100 is the best score and 0 is the worst.
Range of Motion | through study completion, an average of 6 weeks
  the flexion and extension range of motion in degrees of the patient recorded using a goniometer by the physical therapist while in the hospital and surgeon while in the clinic for follow up visits. Normal range of motion is 0-120 degrees.

CONTACTS AND LOCATIONS:
Overall Officials: John W Mann, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Institute for Orthopaedics & Neurosciences, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lund J, Jenstrup MT, Jaeger P, Sorensen AM, Dahl JB. Continuous adductor-canal-blockade for adjuvant post-operative analgesia after major knee surgery: preliminary results. Acta Anaesthesiol Scand. 2011 Jan;55(1):14-9. doi: 10.1111/j.1399-6576.2010.02333.x. Epub 2010 Oct 29. PMID 21039357
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Kapoor R, Adhikary SD, Siefring C, McQuillan PM. The saphenous nerve and its relationship to the nerve to the vastus medialis in and around the adductor canal: an anatomical study. Acta Anaesthesiol Scand. 2012 Mar;56(3):365-7. doi: 10.1111/j.1399-6576.2011.02645.x. PMID 22335278
- [Background] Pepper AM, North TW, Sunderland AM, Davis JJ. Intraoperative Adductor Canal Block for Augmentation of Periarticular Injection in Total Knee Arthroplasty: A Cadaveric Study. J Arthroplasty. 2016 Sep;31(9):2072-6. doi: 10.1016/j.arth.2016.02.030. Epub 2016 Feb 26. PMID 26996675
- [Background] Kavolus JJ, Sia D, Potter HG, Attarian DE, Lachiewicz PF. Saphenous Nerve Block From Within the Knee Is Feasible for TKA: MRI and Cadaveric Study. Clin Orthop Relat Res. 2018 Jan;476(1):30-36. doi: 10.1007/s11999.0000000000000006. PMID 29529612